CLINICAL TRIAL: NCT01988740
Title: Markers of Oxidative Stress in a Early Week Miscarriage: Ischemia of Modified Albumin
Acronym: IMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Hediye Dagdeviren, md, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2013/87
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: First Trimester Pregnancy; Fetal Heart Activity Absent; Absence of Fetal Pole on Ultrasonographic Examination.
Keywords: Ischemia-modified albumin; Recurrent pregnancy loss; Abnormal placenta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The finding that ischemia-modified albumin (IMA) is increased in pre-eclamptic pregnancy suggests a role for IMA as a potential biomarker for abnormal placental development related to miscarriage.This study was undertaken to evaluate IMA levels in women with recurrent pregnancy loss (RPL).

DETAILED DESCRIPTION:
Ischemia-modified albumin (IMA) measured by the albumin cobalt binding test is a relatively new biomarker in the identification of myocardial ischemia. Experimental studies have shown that pregnancies normally develop in a relatively hypoxic intrauterine environment, and the subsequent reperfusion and oxidative stress is important for physiological trophoblast development. The finding that maternal serum IMA levels are raised so early in pregnancy provides further support for IMA as a potential marker for abnormal placental development that may be related to early pregnancy loss. In this study, we aimed to evaluate maternal circulating IMA levels in women with RPL by comparing them with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* first trimester pregnancy
* absence of fetal cardiac activity
* absence of fetal pole
* history of two or more unexplained first trimester miscarriages
* no live births
* apparently healthy women attending for antenatal care in the first trimester with at least one previous uneventful natural pregnancy

Exclusion Criteria:

* pre-existing diabetes or vascular disease were excluded
* diagnosis of chromosomal, anatomic, endocrinologic and autoimmunologic etiology of recurrent pregnancy loss
* Women with multiple pregnancy
* any major or minor fetal anomaly
* current smokers

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: first trimester pregnancy with absence of fetal cardiac activity
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
first trimester pregnant women | under 14 w gestation
  first trimester pregnancy with absence of fetal cardiac activity or absence of fetal pole on ultrasonographic examination Patients with a history of two or more unexplained first trimester miscarriages and no live births were included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: hüseyin cengiz, md, Study Director — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Cengiz H, Dagdeviren H, Kanawati A, Suzen Caypinar S, Yesil A, Ekin M, Yasar L. Ischemia-modified albumin as an oxidative stress biomarker in early pregnancy loss. J Matern Fetal Neonatal Med. 2016;29(11):1754-7. doi: 10.3109/14767058.2015.1061494. Epub 2015 Jul 2. PMID 26135770